CLINICAL TRIAL: NCT02107404
Title: Randomized, Open-label, Parallel-group, Multi-centre Phase II Clinical Trial With Active Cellular Immunotherapy DCVAC/PCa in Patients With Localized Prostate Cancer After Primary Radical Prostatectomy
Brief Title: Phase II Study of DCVAC/PCa Added After Radical Primary Prostatectomy for Patients With Localized Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SOTIO a.s. (Industry)
Responsible Party: Sponsor
Organization: Sotio Biotech Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SP003
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2015-06

CONDITIONS: Prostate Cancer
Keywords: Immunotherapy; Prostate Cancer; Biological; Vaccine
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DCVAC/PCa Arm (Experimental): Dendritic Cells DCVAC/PCA Experimental therapy
  Interventions: Biological: Dendritic Cells DCVAC/PCa
- Standard Therapy (No Intervention): No Intervention

INTERVENTIONS:
Biological: Dendritic Cells DCVAC/PCa — DCVAC/PCa Experimental therapy
  Arms: DCVAC/PCa Arm

SUMMARY:
The purpose of this study is to determine whether DCVAC/PCa added after radical primary prostatectomy can improve PSA doubling times for patients with localized Prostate Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male 18 years and older
* Histologically confirmed pT2 prostate cancer
* Post radical prostatectomy
* PSA values measured after the value greater than 0.020 ng/mL resulted in PSA doubling time (PSADT) equal or less than 12 months
* Salvage radiotherapy naïve with PSA increase within 2 years or after salvage radiotherapy with PSA not higher than 1 ng/ml
* Eastern Cooperative Oncology Group (ECOG) 0-2

Exclusion Criteria:

* Confirmed brain and/or leptomeningeal metastases
* Prior androgen deprivation therapy or orchiectomy for prostate cancer
* Peripheral neuropathy of Common Toxicity Criteria (CTC) grade 2 or greater
* Other uncontrolled intercurrent illness
* Treatment with immunotherapy against prostate cancer
* Clinically significant cardiovascular disease
* Active autoimmune disease requiring treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-04 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2017-05-22 (Actual)

PRIMARY OUTCOMES:
Change in Prostate Specific Antigen (PSA) Doubling Time from randomization to week 40 | 40 Weeks

SECONDARY OUTCOMES:
Change in PSA Doubling Time during Follow-up from week 40 to 2 years after randomization | 104 Weeks
Frequency of Adverse Events | 0, 2, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 52, 65, 78, 91, 104 weeks
Proportion of Patients with Objective disease progression within 2 years | 104 Weeks
Number of Patients requiring further therapy at 2 years | 104 Weeks
Comparison of PSA Doubling Time in Treatment Phase with Immunotherapy with the Value Prior to Randomization | 104 Weeks
Proportion of patients after RPE with biochemical relapse within 2 years of randomization | 104 Weeks
Proportion of patients with progressive increase in PSA within 2 years of randomization | 104 Weeks
Overall survival | 104 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Scheiner, PhD, Study Director — Sotio Accord
Locations (11):
- Czechia (11):
  - Brno
  - Hradec Králové
  - Jablonec nad Nisou
  - Jihlava
  - Mníšek pod Brdy
  - Nový Jičín
  - Olomouc
  - Pilsen
  - Prague
  - Uherské Hradiště
  - Ústí nad Labem